CLINICAL TRIAL: NCT06805773
Title: Evaluating the Use of Educational Videos in a Medical Oncology Sarcoma Clinic to Improve Patient Knowledge and Satisfaction.
Brief Title: Evaluating the Use of Educational Videos in Newly Diagnosed Patients in a Medical Oncology Sarcoma Clinic
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 4693
Record Dates: First submitted 2025-01-23; First posted 2025-02-03 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-01

CONDITIONS: Sarcoma
Keywords: Education; Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Educational Videos (Experimental)
  Interventions: Other: Educational videos
- Standard of Care (Other)
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Educational videos — Participants will be provided with four educational videos in clinic prior to their initial medical oncology consult.
  Arms: Educational Videos
Other: Standard of Care — Participants in the control arm will be provided with the educational videos after their consult with the medical oncologist.
  Arms: Standard of Care

SUMMARY:
This study aims to evaluate how sarcoma-specific educational videos improve patients' knowledge of their disease and treatment options before their first clinic appointment.

Participants will watch four educational videos before their first appointment with a medical oncologist. Participants will be asked to complete surveys to assess their understanding of sarcoma and its treatment options before and after their first medical oncology clinic appointment.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written and voluntary informed consent.
2. Have histologically documented advanced metastatic sarcoma, or is a caregiver of a patient with histologically documented advanced metastatic sarcoma.
3. Age ≥ 18 years.
4. Have not received any previous systemic treatment for sarcoma, or is a caregiver of a sarcoma patient who has not received any previous systemic treatment for sarcoma.
5. Willing/able to complete questionnaires.
6. Able to read and write in English.

Exclusion Criteria:

1. Inability to provide informed consent.
2. Previously seen by a medical oncologist for their sarcoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Assess differences in patients' and caregivers' knowledge and perceptions of sarcoma and its treatment before and after educational intervention | up to 2 weeks (date when given appointment and date of first appointment)
  Evaluate the changes in global responses between baseline surveys and post educational intervention surveys.

SECONDARY OUTCOMES:
Assess understandability and actionability of sarcoma educational videos. | up to 2 weeks (date when given appointment and date of first appointment)
  The Patient Education Materials Assessment Tool (PEMAT) for Audiovisual Materials will be used to assess the video's understandability and actionability. The higher the score (>80%), the more understandable or actionable the material.
Assess understandability and actionability of sarcoma educational videos. | up to 2 weeks (date when given appointment and date of first appointment)
  The Suitability Assessment of Materials (SAM) will be used for evaluation of health-related information for adults to objectively assess the suitability of these educational materials for sarcoma patients.
Assess patient's and caregivers' satisfaction with the educational videos | up to 2 weeks (date when given appointment and date of first appointment)
  Based on responses from a post-educational intervention survey. The scores will be measured using a Likert Scale (1-5), with higher scores indicating greater satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Only IPD used in the results publication will be shared.